CLINICAL TRIAL: NCT01900392
Title: A Randomized Trial of Financial Incentives for Maintenance of Weight Loss
Brief Title: Financial Incentives for Maintenance of Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Duke University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 816917; 1R01AG045045-01 (NIH)
Record Dates: First submitted 2013-06-26; First posted 2013-07-16 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Arm (No Intervention): No other financial incentive other than for the 3-, 6-, 9-, & 12-month weigh-ins and surveys. Participants will receive daily feedback for months 1-6 and will be observed without intervention in Phase II (months 7-12). Two weigh-ins will be required during Phase II, one at 9 months and the other at 12 months.
- Direct payment (Experimental): In addition to the incentives for the 3-, 6-, 9-, & 12-month weigh-ins, participants who meet their daily goal will be eligible to receive an incentive for each day their goal is met during the first 6 months of the study. All daily incentive earnings will be paid out after verifying participants' weights during an in person weigh in at a Weight Watchers location at months 3 and 6. Winnings will be proportional to weight loss. For example, if a participant's goal was to lose 6 pounds by month 3, but he/she only lost 3 pounds, that participant would only receive 50% of their total eligible winnings.
  Similar to the control arm, participants will receive daily feedback for months 1-6 and will be observed without intervention in Phase II (months 7-12). The weigh-ins at 9- and 12-months will also be required.
  Interventions: Behavioral: Financial incentive
- Lottery (Experimental): In addition to the incentives for the 3-, 6-, 9-, & 12-month weigh-ins, participants who meet their daily goal will be eligible for the daily lottery during the first 6 months of the study. The expected daily winning for the lottery is the same as for the direct payment arm. All daily incentive earnings will be paid out after verifying participants' weights during an in person weigh in at a Weight Watchers location at months 3 and 6. Winnings will be proportional to weight loss. For example, if a participant's goal was to lose 6 pounds by month 3, but he/she only lost 3 pounds, that participant would only receive 50% of their total eligible winnings.
  Similar to the control arm, participants will receive daily feedback for months 1-6 and will be observed without intervention in Phase II (months 7-12). The weigh-ins at 9- and 12-months will also be required.
  Interventions: Behavioral: Financial incentive

INTERVENTIONS:
Behavioral: Financial incentive — Participants in the direct payment and lottery arms will receive financial incentives as part of the intervention. See arm descriptions for more detail.
  Arms: Direct payment; Lottery

SUMMARY:
This study aims to evaluate the effectiveness of financial incentives in improving and maintaining weight loss.

DETAILED DESCRIPTION:
Study participants will be obese volunteers recruited from a major community-based weight loss program (Weight Watchers), who have lost at least 5kg during the 4-6 months prior to enrolling in the study. Among these participants, the following will be assessed: 1. The effectiveness of a daily lottery-based financial incentive, relative to the control group, on weight loss and weight maintenance; 2. The effectiveness of a direct payment incentive, relative to the control group, on maintenance of weight loss; 3. Assess the comparative effectiveness of lottery-based and direct payment financial incentives on weight loss and maintenance; 4. The degree to which weight loss is maintained in the intervention groups relative to usual care during the 6 months following cessation of the intervention will also be determined.

During Phase I, incentives will be provided to some study participants (direct payment and lottery arm) for the first 6 months and subjects will be followed for 6 more months to examine effects following cessation of incentives.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 30-80
* BMI between 30 and 45 prior to starting Weight Watchers
* Have a documented weight loss of at least 5kg in the past 4-6 months before enrolling
* Stable health

Exclusion Criteria:

* Substance abuse
* Bulimia nervosa or related behaviors
* Pregnancy or breast feeding
* Medical contraindications to counseling about diet, physical activity, or weight reduction
* Unstable mental illness
* Screen positive for pathological gambling on the basis of the 10 item DSM-IV criteria (excluded if meets 5 or more criteria)
* Individuals unable to read consent forms or fill out surveys in English

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults--The Evidence Report. National Institutes of Health. Obes Res. 1998 Sep;6 Suppl 2:51S-209S. No abstract available. PMID 9813653
- [Background] Office of the Surgeon General (US); Office of Disease Prevention and Health Promotion (US); Centers for Disease Control and Prevention (US); National Institutes of Health (US). The Surgeon General's Call To Action To Prevent and Decrease Overweight and Obesity. Rockville (MD): Office of the Surgeon General (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK44206/ PMID 20669513
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Adams KF, Schatzkin A, Harris TB, Kipnis V, Mouw T, Ballard-Barbash R, Hollenbeck A, Leitzmann MF. Overweight, obesity, and mortality in a large prospective cohort of persons 50 to 71 years old. N Engl J Med. 2006 Aug 24;355(8):763-78. doi: 10.1056/NEJMoa055643. Epub 2006 Aug 22. PMID 16926275
- [Background] Yan LL, Daviglus ML, Liu K, Stamler J, Wang R, Pirzada A, Garside DB, Dyer AR, Van Horn L, Liao Y, Fries JF, Greenland P. Midlife body mass index and hospitalization and mortality in older age. JAMA. 2006 Jan 11;295(2):190-8. doi: 10.1001/jama.295.2.190. PMID 16403931
- [Background] Daviglus ML, Liu K, Yan LL, Pirzada A, Manheim L, Manning W, Garside DB, Wang R, Dyer AR, Greenland P, Stamler J. Relation of body mass index in young adulthood and middle age to Medicare expenditures in older age. JAMA. 2004 Dec 8;292(22):2743-9. doi: 10.1001/jama.292.22.2743. PMID 15585734
- [Background] Finkelstein EA, Trogdon JG, Brown DS, Allaire BT, Dellea PS, Kamal-Bahl SJ. The lifetime medical cost burden of overweight and obesity: implications for obesity prevention. Obesity (Silver Spring). 2008 Aug;16(8):1843-8. doi: 10.1038/oby.2008.290. Epub 2008 May 29. PMID 18535543
- [Background] Nordmann AJ, Nordmann A, Briel M, Keller U, Yancy WS Jr, Brehm BJ, Bucher HC. Effects of low-carbohydrate vs low-fat diets on weight loss and cardiovascular risk factors: a meta-analysis of randomized controlled trials. Arch Intern Med. 2006 Feb 13;166(3):285-93. doi: 10.1001/archinte.166.3.285. PMID 16476868
- [Background] Gardner CD, Kiazand A, Alhassan S, Kim S, Stafford RS, Balise RR, Kraemer HC, King AC. Comparison of the Atkins, Zone, Ornish, and LEARN diets for change in weight and related risk factors among overweight premenopausal women: the A TO Z Weight Loss Study: a randomized trial. JAMA. 2007 Mar 7;297(9):969-77. doi: 10.1001/jama.297.9.969. PMID 17341711
- [Background] Methods for voluntary weight loss and control. NIH Technology Assessment Conference Panel. Consensus Development Conference, 30 March to 1 April 1992. Ann Intern Med. 1993 Oct 1;119(7 Pt 2):764-70. PMID 8363212
- [Background] Giuffrida A, Torgerson DJ. Should we pay the patient? Review of financial incentives to enhance patient compliance. BMJ. 1997 Sep 20;315(7110):703-7. doi: 10.1136/bmj.315.7110.703. PMID 9314754
- [Background] Kane RL, Johnson PE, Town RJ, Butler M. A structured review of the effect of economic incentives on consumers' preventive behavior. Am J Prev Med. 2004 Nov;27(4):327-52. doi: 10.1016/j.amepre.2004.07.002. PMID 15488364
- [Background] Volpp KG, Gurmankin Levy A, Asch DA, Berlin JA, Murphy JJ, Gomez A, Sox H, Zhu J, Lerman C. A randomized controlled trial of financial incentives for smoking cessation. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):12-8. doi: 10.1158/1055-9965.EPI-05-0314. PMID 16434580
- [Background] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Flegal KM, Graubard BI, Williamson DF, Gail MH. Excess deaths associated with underweight, overweight, and obesity. JAMA. 2005 Apr 20;293(15):1861-7. doi: 10.1001/jama.293.15.1861. PMID 15840860
- [Background] Must A, Spadano J, Coakley EH, Field AE, Colditz G, Dietz WH. The disease burden associated with overweight and obesity. JAMA. 1999 Oct 27;282(16):1523-9. doi: 10.1001/jama.282.16.1523. PMID 10546691
- [Background] The sixth report of the Joint National Committee on prevention, detection, evaluation, and treatment of high blood pressure. Arch Intern Med. 1997 Nov 24;157(21):2413-46. doi: 10.1001/archinte.157.21.2413. PMID 9385294
- [Background] Eckel RH. Obesity and heart disease: a statement for healthcare professionals from the Nutrition Committee, American Heart Association. Circulation. 1997 Nov 4;96(9):3248-50. doi: 10.1161/01.cir.96.9.3248. No abstract available. PMID 9386201
- [Derived] Yancy WS Jr, Shaw PA, Reale C, Hilbert V, Yan J, Zhu J, Troxel AB, Foster GD, Volpp KG. Effect of Escalating Financial Incentive Rewards on Maintenance of Weight Loss: A Randomized Clinical Trial. JAMA Netw Open. 2019 Nov 1;2(11):e1914393. doi: 10.1001/jamanetworkopen.2019.14393. PMID 31675083

RESULTS

PARTICIPANT FLOW:
Groups:
- Direct Payment: In addition to the incentives for the 3-, 6-, 9-, & 12-month weigh-ins, participants who meet their daily goal will be eligible to receive an incentive for each day their goal is met during the first 6 months of the study. All daily incentive earnings will be paid out after verifying participants' weights during an in person weigh in at a Weight Watchers location at months 3 and 6. Winnings will be proportional to weight loss. For example, if a participant's goal was to lose 6 pounds by month 3, but he/she only lost 3 pounds, that participant would only receive 50% of their total eligible winnings.
  Similar to the control arm, participants will receive daily feedback for months 1-6 and will be observed without intervention in Phase II (months 7-12). The weigh-ins at 9- and 12-months will also be required.
  Financial incentive: Participants in the direct payment and lottery arms will receive financial incentives as part of the intervention. See arm descriptions for more detail.
Period: Overall Study
Arm/Group | Control Arm | Direct Payment | Lottery
Started | 39 | 75 | 77
Completed | 38 | 74 | 77
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Direct Payment: In addition to the incentives for the 3-, 6-, 9-, & 12-month weigh-ins, participants who meet their daily goal will be eligible to receive an incentive for each day their goal is met during the first 6 months of the study. All daily incentive earnings will be paid out after verifying participants' weights during an in person weigh in at a Weight Watchers location at months 3 and 6. Winnings will be proportional to weight loss. For example, if a participant's goal was to lose 6 pounds by month 3, but he/she only lost 3 pounds, that participant would only receive 50% of their total eligible winnings.
- Control: No other financial incentive other than for the 3-, 6-, 9-, & 12-month weigh-ins and surveys. Participants will receive daily feedback for months 1-6 and will be observed without intervention in Phase II (months 7-12). Two weigh-ins will be required during Phase II, one at 9 months and the other at 12 months.
- Total: Total of all reporting groups
Arm/Group | Lottery | Direct Payment | Control | Total
Number analyzed (Participants) | 77 | 75 | 39 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (10.3) | 48.6 (11.0) | 50.1 (10.0) | 49.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 69 | 36 | 175
  Male | 7 | 6 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 2 | 8
  Not Hispanic or Latino | 75 | 71 | 37 | 183
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 1 | 8
  White | 68 | 69 | 33 | 170
  More than one race | 3 | 1 | 3 | 7
  Unknown or Not Reported | 1 | 1 | 2 | 4
Household income [Count of Participants; unit: Participants]
  <US $50,000 | 12 | 5 | 6 | 23
  US $50,000 to <US $100,000 | 36 | 40 | 20 | 96
  ≥US $100,000 | 29 | 30 | 13 | 72
Household size [Mean (Standard Deviation); unit: people per household] | 3.2 (1.5) | 3.0 (1.4) | 3.0 (1.2) | 3.1 (1.4)
Education [Number; unit: participants]
  Less than college | 26 | 35 | 11 | 72
  College graduate | 28 | 11 | 16 | 55
  Post-college degree | 23 | 29 | 12 | 64
Weight measures [Mean (Standard Deviation); unit: Kilograms]
  Weight at the start of Weight Watchers | 100.8 (15.7) | 101.7 (16.0) | 102.9 (15.6) | 101.6 (15.7)
  Weight at randomization | 89.2 (14.3) | 90.7 (15.7) | 91.2 (15.0) | 90.2 (14.9)
  Weight loss prior to randomization | 11.6 (4.4) | 10.9 (5.1) | 11.7 (4.3) | 11.4 (4.7)
BMI measures [Mean (Standard Deviation); unit: kg/m^2]
  BMI at start of Weight Watchers | 36.5 (4.4) | 36.8 (4.1) | 36.9 (4.5) | 36.7 (4.3)
  BMI at randomization | 32.3 (4.1) | 32.8 (4.3) | 32.6 (4.1) | 32.5 (4.1)
BMI ≥35 kg/m2 at randomization [Count of Participants; unit: Participants] | 26 | 29 | 14 | 69
Eating behaviors by Three-Factor Eating Questionnaire [Mean (Standard Deviation); unit: Scores on a scale] — The raw eating scale scores are transformed to a 0-100 scale [((raw score - lowest possible raw score)/possible raw score range) × 100] Higher scores in the respective scales are indicative of greater cognitive restraint, uncontrolled, or emotional eating
  Scores on a scale
    Cognitive restraint scale | 62.0 (15.0) | 62.6 (14.6) | 62.4 (12.8) | 62.3 (14.4)
    Uncontrolled eating scale | 44.4 (15.6) | 47.6 (16.2) | 41.8 (16.1) | 45.1 (16.0)
    Emotional eating scale | 58.7 (23.8) | 63.3 (23.5) | 55.8 (27.2) | 59.9 (24.5)
Physical activity in min per week [Median (Inter-Quartile Range); unit: Minutes]
  Moderate-vigorous activity min per week | 345 [180 to 885] | 240 [60 to 585] | 390 [180 to 630] | 333 [120 to 700]
  Walking min per week | 180 [53 to 537.5] | 100 [20 to 360] | 150 [90 to 325] | 148 [45 to 428]
  Total activity min per week | 533 [283 to 1295] | 460 [150 to 990] | 600 [270 to 925] | 510 [238 to 1148]

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight From Baseline to 6 Months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Control Arm | Direct Payment | Lottery
Number analyzed (Participants) | 38 | 74 | 77
kilograms | -1.4 (5.8) | -2.8 (5.8) | -3.0 (5.8)
Statistical Analysis 1: Comparison: Control Arm vs Direct Payment vs Lottery; Test type: Other; p > 0.1, Regression, Linear

2. Primary Outcome: Change in Weight From Baseline to 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Control Arm | Direct Payment | Lottery
Number analyzed (Participants) | 38 | 74 | 77
kilograms | 2.8 (16.9) | -2.2 (16.2) | -2.0 (17.9)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Lottery | Direct Payment | Control
All-Cause Mortality (participants affected / at risk) | 0/77 | 1/75 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/77 | 9/75 | 4/39
Other Adverse Events (participants affected / at risk) | 2/77 | 1/75 | 1/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lottery (N=77) | Direct Payment (N=75) | Control (N=39)
Hysterectomy (Reproductive system and breast disorders) | 1 | 1 | 0
Hip replacement (Surgical and medical procedures) | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Brain aneurysm (Nervous system disorders) | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Ruptured appendix (Gastrointestinal disorders) | 0 | 1 | 0
Temporal artery biopsy (Surgical and medical procedures) | 0 | 1 | 0
Lymphoma (Vascular disorders) | 0 | 1 | 0
Syncope (Cardiac disorders) | 0 | 1 | 0
Angina (Cardiac disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Breast cancer (Reproductive system and breast disorders) | 0 | 1 | 0
Vascular surgery (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lottery (N=77) | Direct Payment (N=75) | Control (N=39)
Ganglion cyst outpatient surgery (Surgical and medical procedures) | 0 | 0 | 1
Sciatica from car accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Broken foot (Injury, poisoning and procedural complications) | 1 | 0 | 0
Torn ACL and MCL, broken ankle (Injury, poisoning and procedural complications) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No